CLINICAL TRIAL: NCT02942355
Title: Pilot Trial of Anastrozole and Palbociclib as First-Line Therapy and as Maintenance Therapy After First Line Chemotherapy in Hormone Receptor Positive, HER2-Negative Postmenopausal Metastatic Breast Cancer
Brief Title: Trial of Anastrozole and Palbociclib in Metastatic HER2-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Pfizer (Industry); Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081369; 00017766 (Other: IRB); LCI-BRE-H2N-ANPA-001 (Other: Atrium Health)
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Female Breast Carcinoma; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A: First-line therapy (Experimental): Anastrozole by mouth daily and palbociclib by mouth Days 1-21 on a 28 day cycle
  Interventions: Drug: anastrozole; Drug: Palbociclib
- Cohort B: Maintenance therapy (Experimental): Anastrozole by mouth daily and palbociclib by mouth Days 1-21 on a 28 day cycle
  Interventions: Drug: anastrozole; Drug: Palbociclib

INTERVENTIONS:
Drug: anastrozole — Anastrozole by mouth daily
  Other Names: Arimidex
Drug: Palbociclib — Palbociclib by mouth daily days 1-21 every 28 days
  Other Names: Ibrance

SUMMARY:
This is an open-label, pilot study designed to evaluate the safety and feasibility of combining anastrozole and palbociclib in the following two cohorts: Cohort A) as first-line therapy and Cohort B) as maintenance therapy after first-line chemotherapy in postmenopausal patients with HR-positive, HER2-negative metastatic breast cancer. Pre- and perimenopausal women must receive therapy with an LHRH agonist. The LHRH agonist will be by choice for an approved LHRH agonist administered according to its respective prescribing information. Following informed consent and eligibility check, subjects will be enrolled to either Cohort A or Cohort B.

DETAILED DESCRIPTION:
A total of 40 subjects will be enrolled over an enrollment period of 18-24 months. The study is planned to enroll up to 25 patients in Cohort A (upfront) and 15 patients in Cohort B (maintenance). Subjects will be recruited through Levine Cancer Institute locations and through referrals. Women of any race or ethnic origin who meet the study criteria may participate in this clinical trial. Males will not be eligible for this study. Breast cancer in men is rare and the efficacy of aromatase inhibitors in males is limited. Children are not included in this clinical trial because the effects of palbociclib are not known in the pediatric population, but may be eligible for other pediatric trials.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older, who are either:
* Postmenopausal, as defined by at least one of the following criteria:

  * Age greater than or equal to 60 years;
  * Age less than 60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause and serum estradiol, FSH and LH level within the laboratory reference range for postmenopausal females;
  * Documented bilateral oophorectomy;
  * Medically confirmed ovarian failure OR premenopausal or perimenopausal, i.e., not meeting the criteria for being postmenopausal.
* Premenopausal or perimenopausal women can be enrolled if amenable to be treated with an LHRH agonist. Patients must have commenced treatment with an LHRH agonist at least 4 weeks prior to start of study treatment.
* Histologically or cytological confirmed diagnosis of breast cancer with evidence of metastatic disease. Locally advanced disease not amenable to resection is eligible.
* Documentation of ER-positive and, or PR-positive tumor based on most recent tumor biopsy (unless bone-only disease). ER and PR assays are considered positive if there is at least 1 percent positive in the tumor sample.
* Documentation of HER2-negative tumor based on most recent tumor biopsy. Tumor must not demonstrate overexpression of HER2 by either IHC (immunohistochemistry) or in-situ hybridization (ISH).
* No previous treatment for metastatic disease for Cohort A.

  * For Cohort A: previous treatment with endocrine therapy in the adjuvant or neoadjuvant setting is allowed
  * For Cohort B: only first-line chemotherapy (can be single-agent or a combination regimen) for metastatic disease with response (defined as a complete response or partial response by RECIST version 1.1, or stable disease for six months or more from this regimen) and chemotherapy discontinued for 21 days is allowed; patients may have received prior systemic therapy in the adjuvant or neoadjuvant setting.
* For Cohort A, measurable disease as defined by RECIST version 1.1, or bone-only disease prior to start of study treatment. Patients with bone-only metastatic cancer must have a lytic or mixed lytic-blastic lesion that can be accurately assessed by CT or MRI. Patients with bone-only disease who have blastic-only metastasis are not eligible. Tumor lesions previously irradiated or subjected to other loco regional therapy will only be deemed measurable if progression at the treated site after completion of therapy is clearly documented. For Cohort B, measurable disease as defined by RECIST version 1.1, or evaluable disease.
* Patient has archival tumor tissue available that is formalin-fixed and paraffin-embedded. Biopsy sample taken at the time of presentation with recurrent or metastatic disease is recommended.For patients who do not have archival tissue, tissue from a fresh biopsy should be obtained prior to study treatment initiation, if it can be safely attained using local anesthesia only. One exception is those patients with bone-only disease for whom provision of previous archival tissue would be acceptable. Serial fresh tumor tissue samples will be collected in patients with lesions amenable for a biopsy who consent to such a procedure.
* ECOG performance status 0, 1 or 2.
* Must have normal organ and marrow function as defined below:

  * Hematologic: Absolute neutrophil count greater than or equal to 1,500/mcL;
  * Platelets greater than or equal to 100,000/mcL; Hemoglobin greater than or equal to 9 g/dL.
  * Renal: Serum creatinine less than or equal to 1.5X ULN or Measured or calculated creatinine clearance (CrCl) greater than or equal to 60 mL/min for subject with creatinine levels > 1.5X ULN [CrCl should be calculated per institutional standard; GFR can also be used in place of creatinine or CrCl]
  * Hepatic: Total bilirubin less than or equal to 1.5X ULN; AST(SGOT)/ALT(SGPT) less than or equal to 3X ULN (less than or equal to 5X ULN if liver metastases present); Alkaline phosphatase less than or equal to 2.5X ULN (less than or equal to 5X ULN if liver or bone metastases present)
* Able to swallow and retain oral medication per the Investigator.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with any CDK inhibitor
* Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
* Use of food or drugs known to be potent CYP3A4 inhibitors and drugs known to be potent CYP3A4 inducers (for examples, see the Prohibited Medications Section)
* Major surgery, chemotherapy, radiotherapy, or other anti-cancer therapy within 3 weeks before treatment.
* Any of the following within 6 months prior to study consent: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE Grade 2 or more, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
* Impairment of gastro-intestinal function or GI disease that may significantly alter the absorption of palbociclib, such as history of GI surgery which may result in intestinal blind loops and patients with clinically significant gastroparesis, short bowel syndrome, unresolved nausea, vomiting, active inflammatory bowel disease or diarrhea of CTCAE Grade > 1.
* Prior hematopoietic stem cell or bone marrow transplantation.
* Known hypersensitivity to anastrozole.
* Known human immunodeficiency virus infection.
* Other severe acute or chronic medical or psychiatric condition, that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
* Participation in other studies involving investigational drug(s) within 4 weeks before treatment initiation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with neutropenia that leads to permanent treatment discontinuation | From enrollment to treatment discontinuation; participants remain on treatment until disease progression, unacceptable toxicity, participant withdrawal, or investigator decision. Assessed for approximately 4 years.
  Determined for each subject as a binary variable indicating whether or not the participant experienced any neutropenic adverse event (according to NCI Common Terminology for Adverse Events version 4.0) that leads to permanent treatment discontinuation

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of treatment start to date of death, or censored as described; assessed for approximately 4 years
  Defined as the duration from start of first line metastatic chemotherapy to the date of death from any cause. Participants who are alive or lost to follow up at the time of the analysis will be censored at the last known date they were alive.
Progression Free Survival (PFS) | From treatment start date to date of progression/death, or censored as described; assessed for approximately 4 years.
  PFS is defined as the duration of time from the start of first line metastatic chemotherapy to first occurrence of either progressive disease (PD) or death. PD must be objectively determined per RECIST 1.1 criteria, where progression date is date of the radiologic assessment that identified PD. If subject died without documented PD, progression date will be death date. For surviving subjects who do not have PD, PFS will be censored at the date of last disease assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, PFS will be censored at the date of last disease assessment prior to commencement of subsequent therapy. Subjects who have an initial PFS event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Number of participants with an objective response | From enrollment to best response while on study treatment; participants remain on treatment until disease progression, unacceptable toxicity, participant withdrawal, or investigator decision. Assessed for approximately 4 years.
  Objective response will be determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of complete response (CR) or partial response (PR) as determined by RECIST 1.1 response criteria. A CR is indicated by disappearance of all target and non target lesions. A PR is indicated by >=30% decrease in sum of longest diameter of target lesions with baseline as reference.
Number of participants with clinical benefit | From enrollment to best response while on study treatment; participants remain on treatment until disease progression, unacceptable toxicity, participant withdrawal, or investigator decision. Assessed for approximately 4 years.
  Clinical benefit will be determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of complete response (CR), partial response (PR), or stable disease (SD) for >=6 months as determined by RECIST 1.1 response criteria. A CR is indicated by disappearance of all target and non target lesions. A PR is indicated by >=30% decrease in sum of longest diameter of target lesions with baseline as reference. SD is indicated by neither sufficient shrinkage to qualify for PR nor sufficient growth from nadir (>=20%) to indicate progression.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Tan, MD, Principal Investigator — Atrium Health (formerly Carolinas HealthCare System)
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study of aromatase inhibitor and palbociclib in HR+HER2-negative metastatic breast cancer — https://www.ncbi.nlm.nih.gov/pubmed/27959613

DOCUMENTS (1):
  • Informed Consent Form (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT02942355/ICF_000.pdf